CLINICAL TRIAL: NCT05690243
Title: Minds Navigating the Diagnosis of Mild Cognitive Impairment (MiND-MCI)
Brief Title: Minds Navigating the Diagnosis of Mild Cognitive Impairment
Acronym: MIND-MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lori Davis, MD, Associate Chief of Staff, Research Service, Tuscaloosa Veterans Affairs Medical Center, Tuscaloosa Research & Education Advancement Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170
Record Dates: First submitted 2022-11-21; First posted 2023-01-19 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Cognitive Dysfunction; Mild Cognitive Impairment
Keywords: therapy; video telehealth; veteran
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: two-arm, single-blind, pilot randomized controlled trial with 1:1 randomization. Wait List Control.
Who Masked: Outcomes Assessor
Masking Description: Assessor and fidelity monitor will be blinded to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group therapy delivered via video telehealth (Experimental): Nine sessions of 60 min each group therapy delivered via telehealth
  Interventions: Behavioral: Group psychotherapy delivered via video telehealth
- Group therapy delivered via video telehealth - wait list control (Other): Nine sessions of 60 min each group therapy delivered via telehealth after a waiting period.
  Interventions: Behavioral: Group psychotherapy delivered via video telehealth

INTERVENTIONS:
Behavioral: Group psychotherapy delivered via video telehealth — Small group psychotherapy using psychoeducation and skills training aimed at addressing modifiable factors in MCI.

SUMMARY:
The goal of this clinical trial is to find out if a 9 week group therapy using video from home will help veterans with Mild Cognitive Impairment (MCI). The main questions it aims to answer are:

* is the video therapy user-friendly for veterans?
* does it improve veterans well-being and quality-of-life?

Veterans will be asked to attend nine 1 hour small group video sessions and will complete questionnaires before and after the sessions.

Researchers will compare the group of veterans that starts the video sessions right away with a group that waits before starting the video sessions.

DETAILED DESCRIPTION:
The study will be achieved by conducting a two-arm, single-blind, pilot randomized controlled trial at two VA medical centers. Eighty participants at each site will be randomized in a 1:1 ratio to either the MiND-MCI group or waitlist control group. Participants will be Veterans ages 60 and older with a diagnosis of MCI, at least one cardiovascular risk factor, self-reported cognitive complaint, and self-reported difficulty adjusting to MCI diagnosis or symptoms. MiND-MCI will be delivered in nine weekly 60-minute sessions via telehealth in groups of 5 to 7 Veterans. Feasibility and acceptability process data will be tracked throughout the study. Acceptability measures pertaining to participants' perceptions of MiND-MCI will be collected at post-treatment using quantitative and qualitative assessment methods. Outcome measures collected at baseline, post-treatment, and 12-week follow-up will assess global QoL, MCI-related QoL, MCI-related self-efficacy, depression, anxiety, loneliness, coping, and cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* age 60 or older
* diagnosis of MCI, diagnosed at least a month or longer prior to screening
* diagnosis of at least one cardiovascular risk factor (i.e., hypertension, diabetes mellitus II, hyperlipidemia/hypercholesterolemia, or obesity)
* self-reported cognitive complaint (i.e., "Do you have problems with your memory or thinking abilities?")
* self-reported difficulty adjusting to declines in cognitive functioning (i.e., "Have these problems with memory or thinking impacted you, your life, or others in your life?")
* English speaking, and (h) ability to provide written informed consent

Exclusion Criteria:

* diagnosis of dementia or a neurodegenerative disorder
* diagnosis of serious mental illness likely to impact cognition (i.e., schizophrenia or bipolar I disorder)
* acutely suicidal or homicidal
* actively psychotic
* active substance use disorder
* limited life expectancy due to a terminal medical condition
* receiving ongoing chemotherapy or radiation treatment at time of screening
* residing in an assisted living or residential care facility
* currently participating in another psychotherapy, health promotion intervention, or cognitive training program, and
* any significant changes to psychotropic medications or medications for memory and cognition in the past month. Participants prescribed psychotropic medications and medications for memory and cognition will be asked to stay on their current dosages for the duration of the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a group video-telehealth intervention for veterans with MCI | At Week 0 (randomization)
  percentage of screened, eligible subjects that enroll in intervention
Acceptability of a group video-telehealth intervention for veterans with MCI | At Week 10 (one week after completion of the 9 video-telehealth sessions)
  percentage of subjects that attend 70% or more of scheduled sessions

SECONDARY OUTCOMES:
Change in the Quality of Life in Alzheimers Disease (QOL-AD, range of 13-52) scale in Veterans with Mild Cognitive Impairment following participation in a 9-week video-telehealth intervention. | baseline to 12 week post-treatment follow-up visit
  change in the Quality of Life in Alzheimers Disease (QOL-AD) Scale

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Pilkinton, MD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center; Lindsay Jacobs, PhD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Tuscaloosa VA Medical Center, Tuscaloosa, Alabama
  - Salem VA Medical Center, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No